CLINICAL TRIAL: NCT05157321
Title: Effect of Repetitive Transcranial Magnetic Stimulation on Essential Tremors
Brief Title: Repetitive Transcranial Magnetic Stimulation in Essential Tremors Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Fathy Mohammed Mohammed, physician, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0000039
Record Dates: First submitted 2021-12-08; First posted 2021-12-15 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Essential Tremor
Keywords: rTMS, essential tremors
MeSH Terms: conditions — Essential Tremor | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Active Comparator): The patients in this group will receive active repetitive transcranial magnetic stimulation sessions for 4 weeks.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- control group (Sham Comparator): The patients in this group will receive sham repetitive transcranial magnetic stimulation sessions for 4 weeks.
  Interventions: Device: Sham Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — TMS device will deliver repetitive trains of magnetic pulses using Magstim Rapid 2 with angulated figure of eight shaped coil. The device comprised two-channel Neuro-EMG-MS digital system for determining the motor threshold of the patients that will be used for establishing the threshold intensity for stimulation. The figure of eight-shaped coil generated a magnetic field of up to 4 Tesla that penetrates the cranium, enters into the soft tissue of the brain and henceforth stimulates the motor neurons.
  Arms: Study Group
Device: Sham Repetitive Transcranial Magnetic Stimulation — Sham Repetitive Transcranial Magnetic Stimulation
  Arms: control group

SUMMARY:
The aim of the study is to investigate the Effect of Repetitive Transcranial Magnetic Stimulation on Essential Tremors.

DETAILED DESCRIPTION:
Prior to start of rTMS sessions, Clinical evaluation and scaling of tremors using the ET rating scale (Fahn, Tolosa, Marin Tremor Rating Scale) will be employed on the participants in both groups.

rTMS frequency of 1Hz will be delivered to each of the participants in both groups. Each session will be administered once daily for 3 days a week for 4 weeks. 1200 pulses (30 pulses per train with total 40 trains having inter-train delay of 3 seconds) per session will be provided with the coil placed on both cerebellar hemispheres. rTMS frequency of 1Hz was kept constant based on previous studies.

rTMS sessions will be administered by trained professionals who was kept blinded to the research protocols used in the study. After completion of therapeutic programs (after 4 weeks), the participants will be asked to undergo post assessment of Fahn, Tolosa, Marin Tremor Rating Scale at the end of last rTMS session, 1 month, 3 months later.

ELIGIBILITY:
Inclusion Criteria:

1. Patient diagnosed with Essential tremors or Essential tremors plus based on the movement disorders consensus criteria(appendix 1)
2. Patient should have significant residual tremors despite of using appropriate medical treatment.
3. Age: patient should be above 18 years old.
4. Gender: males and females.

Exclusion Criteria:

1. Patients with history of seizures.
2. Patient receiving tremor active drugs including:

   * Central cholinergic drugs (acetylcholine chloride, muscarinic and nicotinic agonists, anticholinesterases, and aminopropranolols)
   * Central monoaminergic drugs (neuroleptics, phenylethylamines, and indoles)
   * Peripheral adrenergic drugs (lithium carbonate, amphetamine sulfate, adrenocorticosteroids, and thyroid hormone supplements)
   * Anticonvulsants (valproic acid), bronchodilators (theophylline and terbutaline sulfate)
   * Antidepressants (amitriptyline hydrochloride).
3. patients who have metal or electronic device implanted in their body such as :

   * cardiac peace maker
   * Aneurysm clips or coils
   * Stents in the neck or brain
   * Deep brain stimulators
   * Spinal cord stimulators
   * Electrodes to monitor brain activity
   * Metallic implants in ears and eyes
   * Bullet fragments in or near the head
   * Baclofen pumps
   * Other metal devices or object implanted in or near the head

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
change in severity of essential tremors | 1 day, 1 month, and 3 months following the end of treatment.
  Fahn, Tolosa, Marin Tremor Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Al-Bahay M. Reda, professor, Study Chair — Faculty of Medicine, Al-Azhar University
Locations (1):
- Al-Azhar university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No